CLINICAL TRIAL: NCT02966548
Title: A Phase 1 Study of the Safety, Tolerability, and Efficacy of Anti-LAG-3 Monoclonal Antibody (BMS-986016) Administered Alone and in Combination With Anti-PD-1 Monoclonal Antibody (Nivolumab, BMS-936558) in Advanced Solid Tumors
Brief Title: Safety Study of BMS-986016 With or Without Nivolumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-034
Record Dates: First submitted 2016-11-01; First posted 2016-11-17 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — relatlimab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monotherapy (Experimental): Relatlimab (BMS-986016) administered every 2 weeks as a single agent intravenous formulation
  Interventions: Drug: Relatlimab
- Combination Therapy (Experimental): Relatlimab (BMS-986016) will be administered in combination with Nivolumab every 2 weeks or every 4 weeks as an intravenous formulation
  Interventions: Drug: Relatlimab; Drug: Nivolumab

INTERVENTIONS:
Drug: Relatlimab — Specified dose on specified days
  Other Names: BMS-986016
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Combination Therapy

SUMMARY:
This study will be used to determine the safety and tolerability of BMS-986016 administered alone and in combination with Nivolumab in subjects with advanced solid tumors.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have histologic or cytologic confirmation of an incurable solid malignancy that is advanced (metastatic and/or unresectable)
* Must have received, and then progressed or been intolerant to, standard treatment regimen in the advanced or metastatic setting, if such a therapy exists
* Presence of at least one lesion with measurable disease as defined by RECIST v1.1 criteria for response assessment
* Males and Females, ages 20 years or older, inclusive

Exclusion Criteria:

* Known or suspected CNS (central nervous system) metastases or with the CNS as the only site of active disease
* Other concomitant malignancies (with some exceptions per protocol)
* Any active autoimmune disease or history of known or suspected autoimmune disease
* History of uncontrolled or significant cardiovascular disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (AE) | Approximately 2.2 years
Number of serious adverse events (SAE) | Approximately 2.2 years
Number of deaths | Approximately 2.2 years
Number of laboratory abnormalities | Approximately 2.2 years

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Time of maximum observed serum concentration (Tmax) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Trough observed serum concentration (Ctrough) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Concentration at the end of a dosing interval (Ctau) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Average concentration over a dosing interval [AUC(TAU)/tau] (Css,avg) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Area under the serum concentration-time curve in 1 dosing interval [AUC(TAU)] of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Total body clearance (CLT) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Volume of distribution at steady state (Vss) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Effective elimination half-life (T-HALFeff) that explains the degree of AUC accumulation observed (T-HALFeff AUC) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Effective elimination half-life that explains the degree of Cmax accumulation observed (T-HALFeff Cmax) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Accumulation index; ration of AUC(TAU) at steady state to AUC(TAU) after the first dose (AI_AUC) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Cmax accumulation index; ratio of Cmax at steady state to Cmax after the first dose (AI_Cmax) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Ctau accumulation index; ratio of Ctau at steady state to Ctau after the first dose (AI_Ctau) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Degree of fluctuation or fluctuation index ([Cmax - Ctau]/Css,avg) (DF) of BMS-986016 | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Best overall response (BOR) | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Duration of response (DOR) | Cycle 1, 2, 3, 4, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Frequency of positive anti-drug antibody (ADA) to BMS-986016 | Cycle 1, 2, 3, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up
Frequency of positive anti-drug antibody (ADA) to Nivolumab | Cycle 1, 2, 3, 5, 9, 13, 17, 21 (28 days/cycle), 60-day follow-up, 135-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Kashiwa-shi, Chiba, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT02966548.html